CLINICAL TRIAL: NCT01606319
Title: Acetaminophen vs. Ibuprofen in Children With Asthma
Brief Title: Acetaminophen Versus Ibuprofen in Children With Asthma
Acronym: AVICA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, dave mauger, Principal Investigator, AsthmaNet Data Coordinating Center, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AsthmaNet 005; 1U10HL098115 (NIH)
Record Dates: First submitted 2012-05-23; First posted 2012-05-25 (Estimated); Results first posted 2017-01-16 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2016-11

CONDITIONS: Asthma; Wheezing
Keywords: Asthma; Wheezing; Ibuprofen; Acetaminophen; exacerbations; pain; fever
MeSH Terms: conditions — Asthma; Respiratory Sounds; Pain; Fever | interventions — Acetaminophen; Ibuprofen; Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- acetaminophen (Experimental): acetaminophen given as needed for pain or fever
  Interventions: Drug: Acetaminophen
- ibuprofen (Experimental): ibuprofen given as needed for pain or fever
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Acetaminophen — 15 mg/kg every 6 hours as needed
  Other Names: tylenol; paracetamol
  Arms: acetaminophen
Drug: Ibuprofen — 9.4 mg/kg every 6 hours as needed
  Other Names: motrin; advil; nonsteroidal anti-inflammatory drug
  Arms: ibuprofen

SUMMARY:
The Acetaminophen Versus Ibuprofen in Children with Asthma study will test the primary hypothesis that in preschool children 12-59 months of age with persistent asthma on standardized asthma therapy, the number of asthma exacerbations requiring systemic corticosteroids will be more frequent in children randomized to receive acetaminophen as compared to those randomized to receive ibuprofen on an as needed basis for fevers and pain.

DETAILED DESCRIPTION:
AVICA is a 48-week randomized therapeutic trial involving two parallel treatment arms: acetaminophen and ibuprofen. Participating children will be randomized to receive either acetaminophen or ibuprofen administered as needed per parental decision for fever and analgesia. This study will address which is the most appropriate antipyretic-analgesic medication in young children with asthma, and will inform both clinicians and parents seeking to treat children with fever and pain. Given the high frequency of administration of these drugs, this study will have a significant impact on pediatric healthcare regardless of whether a differential effect is discovered as significant uncertainty currently exists as to whether acetaminophen use is associated with increased asthma symptoms.

ELIGIBILITY:
Inclusion Criteria:

* 12-59 months of age.
* If the child is not currently taking long-term asthma controller therapy (meaning that the child has taken no inhaled corticosteroid or leukotriene receptor antagonist medication whatsoever over the past 6 months), then one of the following criteria must be met:

  * Daytime asthma symptoms more than two days per week (average over the past 4 weeks),
  * At least one nighttime awakening from asthma (over the past 4 weeks),
  * Two or more asthma exacerbations requiring systemic corticosteroids in the previous 6 months,
  * Four or more wheezing episodes in the previous 12 months.
* If the child is currently taking long-term asthma controller therapy (meaning that the child has taken daily or intermittent/as-needed inhaled corticosteroid or leukotriene receptor antagonist over the past 6 months), then one of the following criteria must be met:

  * Taking inhaled corticosteroid or leukotriene receptor antagonist for more than 3 months (or more than 90 days) out of the previous 6 months (or 180 days),
  * Daytime asthma symptoms more than two days per week (average over the past 4 weeks),
  * More than one nighttime awakening from asthma (over the past 4 weeks),
  * Two or more asthma exacerbations requiring systemic corticosteroids in the previous 12 months,
  * Four or more wheezing episodes in the previous 12 months.
* Up to date with immunizations, including varicella (unless the subject has already had clinical varicella).
* Willingness to provide informed consent by the child's parent or guardian.

Exclusion Criteria:

* Allergic reaction to the study medications or any component of the study drugs, including (but not limited to) urticaria, rash, angioedema, or hypotension following delivery,
* Chronic medical disorders that could interfere with drug metabolism/excretion (for instance chronic hepatic, biliary, or renal disease),
* Chronic medical disorders that may increase the risk of drug-related injury, including (but not limited to):

  * Osteogenesis imperfecta (increased risk of bone demineralization/fracture with corticosteroid therapy),
  * Crohn's disease, ulcerative colitis, juvenile rheumatoid arthritis, clotting disorders, or Factor deficiency (increased risk of bleeding with corticosteroid therapy),
  * G6PD deficiency (increased risk of hemolytic anemia with acetaminophen use),
  * Phenylketonuria (potential for aspartame exposure with study interventions),
  * Seizure disorder treated with anticonvulsants (risk of acetaminophen toxicity with carbamazepine), or
  * History of clotting disorders or Factor deficiency (increased risk of bleeding with corticosteroids),
* Co-morbid disorders associated with wheezing including (but not limited to) immune deficiency disorders, cystic fibrosis, aspiration, clinically-relevant gastroesophageal reflux, tracheomalacia, congenital airway anomalies (clefts, fistulas, slings, rings), bronchiectasis, bronchopulmonary dysplasia, and/or history of premature birth before 35 weeks gestation,
* Significant developmental delay/failure to thrive, defined as 5th percentile for height and/or weight or crossing of two major percentile lines during the last year for age and sex,
* History of a near-fatal asthma exacerbation requiring intubation or assisted ventilation,
* No primary medical caregiver (e.g., a nurse practitioner, physician assistant, physician, or group medical practice such as a hospital-based clinic) whom the subject can contact for primary medical care,
* Three or more hospitalizations in the previous 12 months for wheezing or respiratory illnesses,
* Treatment with 5 or more courses of systemic corticosteroids (oral, intramuscular or intravenous) in the past 6 months,
* Current use of higher than step 2 NAEPP asthma guideline therapy
* If receiving allergy shots, change in the dose within the past 3 months.

Ages: 12 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2013-02; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William B Busse, MD, Study Chair — University of Wisconsin, Madison
Locations (15):
- United States (15):
  - University of Arizona College of Medicine, Tucson, Arizona
  - Children's Hospital & Research Center Oakland, Oakland, California
  - UCSF Benioff Children's Hospital, San Francisco, California
  - National Jewish Health, Denver, Colorado
  - Emory University, Atlanta, Georgia
  - Rush University Medical Center/Stroger Hospital, Chicago, Illinois
  - Children's Memorial Hospital, Chicago, Illinois
  - Children's Hospital Boston, Boston, Massachusetts
  - Children's Hospital, Boston, Boston, Massachusetts
  - St. Louis Children's Hospital, St Louis, Missouri
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Rainbow Babies and Children's Hospital, Case Western Reserve University, Cleveland, Ohio
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - University of Virginia Health System, Charlottesville, Virginia
  - University of Wisconsin-Madison, Madison, Wisconsin

REFERENCES:
- [Derived] Sheehan WJ, Mauger DT, Paul IM, Moy JN, Boehmer SJ, Szefler SJ, Fitzpatrick AM, Jackson DJ, Bacharier LB, Cabana MD, Covar R, Holguin F, Lemanske RF Jr, Martinez FD, Pongracic JA, Beigelman A, Baxi SN, Benson M, Blake K, Chmiel JF, Daines CL, Daines MO, Gaffin JM, Gentile DA, Gower WA, Israel E, Kumar HV, Lang JE, Lazarus SC, Lima JJ, Ly N, Marbin J, Morgan WJ, Myers RE, Olin JT, Peters SP, Raissy HH, Robison RG, Ross K, Sorkness CA, Thyne SM, Wechsler ME, Phipatanakul W; NIH/NHLBI AsthmaNet. Acetaminophen versus Ibuprofen in Young Children with Mild Persistent Asthma. N Engl J Med. 2016 Aug 18;375(7):619-30. doi: 10.1056/NEJMoa1515990. PMID 27532828

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Acetaminophen | Ibuprofen
Started | 150 | 150
Completed | 116 | 110
Not Completed | 34 | 40
Not completed — Lost to Follow-up | 17 | 14
Not completed — Withdrawal by Subject | 9 | 12
Not completed — Physician Decision | 1 | 2
Not completed — Lack of Efficacy | 6 | 8
Not completed — Adverse Event | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acetaminophen | Ibuprofen | Total
Number analyzed (Participants) | 150 | 150 | 300
Age, Continuous [Mean (Standard Deviation); unit: months] | 40.3 (12.9) | 39.4 (13.6) | 39.9 (13.2)
Gender [Count of Participants; unit: Participants]
  Female | 64 | 57 | 121
  Male | 86 | 93 | 179
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 35 | 37 | 72
  Not Hispanic or Latino | 115 | 113 | 228
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 5
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 3 | 0 | 3
  Black or African American | 47 | 50 | 97
  White | 74 | 74 | 148
  More than one race | 22 | 23 | 45
  Unknown or Not Reported | 0 | 0 | 0
Number of urgent care and ED visits in the past year [Mean (Standard Deviation); unit: urgent care/ED visits per year] | 3.1 (2.5) | 3.0 (2.3) | 3.1 (2.4)
Number of Oral Corticosteroid (OCS) courses in the past 6 months [Mean (Standard Deviation); unit: OCS courses per 6 months] | 1 (1.1) | 1.2 (1.0) | 1.1 (1.1)
IgE (kU/L) [Median (Inter-Quartile Range); unit: kU/L] | 64 [19 to 176] | 70 [24 to 252] | 70 [22 to 208]
Allergen Test [Number; unit: participants]
  Positive test | 64 | 62 | 126
  Negative test | 86 | 88 | 174

OUTCOME MEASURES:

1. Primary Outcome: Exacerbation Frequency
Description: the number of asthma exacerbations requiring systemic corticosteroids
Time Frame: last 46 weeks of 48 week treatment period
Population: Two participants in the ibuprofen arm dropped out of the study during the first two weeks of the study and were not included in the analysis per the pre-specified analysis plan.
Measure: Mean (95% Confidence Interval); unit: asthma exacerbations per 46 weeks
Arm/Group | Acetaminophen | Ibuprofen
Number analyzed (Participants) | 150 | 148
asthma exacerbations per 46 weeks | 0.81 [.65 to 1.02] | .87 [.69 to 1.1]
Statistical Analysis 1: Comparison: Acetaminophen vs Ibuprofen; Test type: Superiority or Other; p = 0.67, log-linear model; log-linear model in which the number of exacerbations was assumed to follow a negative binomial distribution; relative rate = 0.94, 95% CI 2-sided [.69 to 1.28] — relative rate with acetaminophen in the numerator and ibuprofen in the denominator

2. Secondary Outcome: Asthma Control Days
Description: proportion of study days on which asthma was controlled, measured by electronic diary
Time Frame: last 46 weeks of 48 week treatment period
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: proportion of days
Arm/Group | Acetaminophen | Ibuprofen
Number analyzed (Participants) | 150 | 148
proportion of days | .86 [.84 to .88] | .87 [.85 to .89]
Statistical Analysis 1: Comparison: Acetaminophen vs Ibuprofen; Test type: Superiority or Other; p = 0.5, ANCOVA; Mean Difference (Final Values) = -.01, 95% CI 2-sided [-0.039 to .0019]

3. Secondary Outcome: Asthma Rescue Medication Use
Description: average albuterol rescue use per week, measured by electronic diary
Time Frame: last 46 weeks of 48 week treatment period
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: inhalations per week
Arm/Group | Acetaminophen | Ibuprofen
Number analyzed (Participants) | 150 | 148
inhalations per week | 2.8 [2.3 to 3.3] | 3 [2.4 to 3.6]
Statistical Analysis 1: Comparison: Acetaminophen vs Ibuprofen; Test type: Superiority or Other; p = 0.69, ANCOVA; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.9 to 0.6]

4. Secondary Outcome: Health Care Utilization
Description: frequency of unscheduled physician visits, emergency department visits or hospitalizations for asthma
Time Frame: last 46 weeks of 48 week treatment period
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: unscheduled health visits per 46 weeks
Arm/Group | Acetaminophen | Ibuprofen
Number analyzed (Participants) | 150 | 148
unscheduled health visits per 46 weeks | .75 [.6 to .95] | .76 [.6 to .97]
Statistical Analysis 1: Comparison: Acetaminophen vs Ibuprofen; Test type: Superiority or Other; p = .94, log-linear model; log-linear model in which the number of exacerbations was assumed to follow a negative binomial distribution; relative rate = 0.99, 95% CI 2-sided [0.72 to 1.37] — relative rate with acetaminophen in the numerator and ibuprofen in the denominator

ADVERSE EVENTS:
Arm/Group | Acetaminophen | Ibuprofen
Serious Adverse Events (participants affected / at risk) | 6/150 | 12/150
Other Adverse Events (participants affected / at risk) | 135/150 | 124/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acetaminophen (N=150) | Ibuprofen (N=150)
asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 8 (8)
Influenza (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Simple laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
tonsilitis (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acetaminophen (N=150) | Ibuprofen (N=150)
Otitis media NOS (Ear and labyrinth disorders) | 37 (56) | 34 (60)
Acute uri (Respiratory, thoracic and mediastinal disorders) | 94 (279) | 73 (198)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 39 (76) | 38 (57)
Strep sore throat (Infections and infestations) | 16 (19) | 13 (14)
Fever (General disorders) | 92 (230) | 75 (176)
Headache (General disorders) | 13 (22) | 15 (33)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 10 (17) | 9 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 32 (55) | 30 (61)
Vomiting (Gastrointestinal disorders) | 17 (18) | 17 (17)
Diarrhea (Gastrointestinal disorders) | 10 (11) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No